CLINICAL TRIAL: NCT06193720
Title: The Impact of Arnica Montana on Postoperative Pain, Swelling and Trismus Following the Surgical Extraction of Impacted Third Molars: A Split Mouth Randomized Clinical Double Blinded Trial
Brief Title: The Impact of Arnica Montana Following the Surgical Extraction of Impacted Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Christian Makary, Professor, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XFMD126
Record Dates: First submitted 2023-12-05; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Edema; Pain; Trismus
MeSH Terms: conditions — Edema; Pain; Trismus | interventions — Arnicae flos extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arnica Montana (Experimental): Patients will take Arnica montana before and after surgery
  Interventions: Drug: Arnica montana
- Control (Placebo Comparator): Patients will take placebo pills to compare the results
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Arnica montana — Assess the effect of arnica montana on pain, swelling ans trismus after impacted third molar surgery
  Arms: Arnica Montana
Other: Placebo — Patients will take placebo drug after surgeries
  Arms: Control

SUMMARY:
Aim: The aim of this study is to evaluate the action of the homeopathic plant Arnica Montana on postoperative edema, pain and trismus after surgical extraction of impacted wisdom teeth.

Materials and Methods: The study is a double-blinded clinical trial recruiting patients undergoing surgical extraction of symmetrically impacted maxillary or mandibular third molars (right and left side). Patients receive alternately and randomly the verum (Arnica Montana 12 CH) or the placebo, in the form of capsules, to be taken 1 day prior to surgery and for 7 days postoperatively. Clinical parameters are collected and include: pain score, maximum mouth opening and facial measurements to assess edema's intensity.

ELIGIBILITY:
Inclusion Criteria:

* Symmetrically impacted bilateral third molars (mandibular or maxillary).
* Young patients aged between 16 and 40 years old.
* No consumption of tobacco or coffee.
* Consent to the terms and conditions of the study.
* Good oral hygiene.
* ASA 1.

Exclusion Criteria:

* Not symmetrically impacted third molars
* Patients with health problems

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Pain VSA | at 0,1,2,3,4,5,6,7 days after surgery
  Assessment of pain on visual analogue scale (between 0 and 10, 0 being no pain at all and 10 being the worst pain)
Amount of face Swelling | at 0,2,7 days after surgery
  Assessment of swelling after the intervention using a flexible ruler to measure the distance between fixed fixed reference points marked on the face:
  * G: Mandibular angle
  * C: External canthus
  * T: Tragus
  * S: Sub-nasal point
  * P: Pogonion
Trismus intensity | at 0,2 and 7 days after surgery
  Assessment of limitation of mouth opening after intervention between the incisal edges of the maxillary and the mandibular central incisors using a vernier caliper

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided